CLINICAL TRIAL: NCT01232517
Title: A Prospective Evaluation of the Dynamic Function of the NeuroVision® System for the Placement of Lumbar Pedicle Screws
Brief Title: NeuroVision® Dynamic Screw Test Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.NV0804
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Spinal Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to gather information about the NeuroVision System (which is FDA cleared for this indication) during the placement of pedicle screws. NeuroVision is a machine that monitors nerve activity during surgery and will alert the surgeon if there are any nerve-related issues during screw placement. The use of nerve monitoring is standard of care at most centers during spine surgery. The standard monitoring for screws placed is performed after the screw is placed, to ensure it is well positioned in the bone (if it is not, the screw may be removed and/or repositioned). The NeuroVision System has a novel feature called "Dynamic Screw Test" that allows for that monitoring to be performed as the screw is placed, rather than after the fact. This study is being done to determine if this real-time monitoring of screw placement provides beneficial additional information to the operating surgeon to prevent misplacement of screws before it happens.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who are at least 18 years of age.
2. Surgical candidates for posterior instrumented lumbar fusion surgery.
3. Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the study.

Exclusion Criteria:

1. Patients with underlying neurological disease or neurological deficits that are not associated with the condition for which they are seeking surgical intervention.
2. Patients who have had previous instrumented surgery at the involved lumbar level.
3. Participants in any other clinical study involving an investigational device or drug within 30 days of enrollment into the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical candidates for posterior instrumented lumbar fusion surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Sensitivities/specificities of NeuroVision Basic and Dynamic Screw Test monitoring modalities to predict (1) pedicle breach and (2) neural injury | 6 weeks postoperative

SECONDARY OUTCOMES:
The change in subject self-reported pain ratings (Visual Analog Scales, leg and back pain) from the preoperative period through postoperative follow-up. | 6 weeks postoperative
Intraoperative time (in minutes) taken to place Basic vs Dynamically tested screws. | Intraoperative
Intraoperative fluoroscopy (in minutes) used to place Basic vs Dynamically tested screws. | Intraoperative

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Northwest Orthopaedic Specialists, PS, Spokane, Washington
  - Aurora BayCare Medical Center, Green Bay, Wisconsin